CLINICAL TRIAL: NCT00969917
Title: A Phase 2, Open-Label Study Evaluating the Efficacy and Safety of IPI 504 in Patients With Advanced Dedifferentiated Liposarcoma
Brief Title: Study Evaluating the Efficacy and Safety of IPI 504 in Patients With Advanced Dedifferentiated Liposarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision not to start the study
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Eduardo Rodenas, MD, Infinity Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-504-09
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Dedifferentiated Liposarcoma
MeSH Terms: conditions — Liposarcoma | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-504 (Experimental): IPI 504 administered twice weekly for 2 weeks followed by 1 week off treatment
  Interventions: Drug: IPI-504

INTERVENTIONS:
Drug: IPI-504 — IPI 504 administered twice weekly at 225 mg/m2 for 2 weeks followed by 1 week off treatment

SUMMARY:
The primary objective of the study is to determine the safety profile and overall response rate of IPI 504 in patients with advanced dedifferentiated liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing informed consent.
* Histologic diagnosis of dedifferentiated liposarcoma.
* Available archival pathology specimen or tissue sample from a new biopsy for confirmation of diagnosis by central pathology reading.
* At least one prior chemotherapy regimen for dedifferentiated liposarcoma.
* No more than 2 prior chemotherapy regimens for dedifferentiated liposarcoma. Note: Any number of non-chemotherapy regimens is permitted.
* Measurable disease on computed tomography (CT) or magnetic resonance imaging (MRI) as defined by RECIST (version 1.1) with at least one measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1.
* Life expectancy ≥6 months.

Exclusion Criteria:

* Prior treatment with any heat shock protein 90 (Hsp90) inhibitor.
* Surgery, radiotherapy, or lesion ablative procedure to the only area of measurable disease
* Patients with prior hepatic resections or hepatic-directed therapy
* Use of a medication or food that is a clinically relevant CYP3A inhibitor or inducer within 2 weeks prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12

PRIMARY OUTCOMES:
To determine the safety profile and overall response rate (ORR) of IPI 504 in patients with advanced dedifferentiated liposarcoma. | Every 6 weeks

SECONDARY OUTCOMES:
To determine the clinical benefit rate and duration of overall response | Every 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States